CLINICAL TRIAL: NCT02524366
Title: A Randomized Study of Transcorporal Versus Standard Artificial Urinary Sphincter Placement
Brief Title: A Study of Transcorporal Versus Standard Artificial Urinary Sphincter Placement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn on November 2017 due to no subject accrual. No subjects were enrolled in this study.
Sponsor: University of Minnesota (Other)
Collaborators: Baylor College of Medicine (Other); University of Iowa (Other); University of Kansas (Other); Loyola University Chicago (Other); Lahey Clinic (Other); University of California, San Francisco (Other); University of Washington (Other); New York University (Other); University of California, San Diego (Other); University of Utah (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Elliott TC vs ST AUS
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; Artificial Urinary Sphincter
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Urinary Sphincter, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcorporal AUS (Experimental): The artificial urinary sphincter is placed through the tunica albuginea of the corpora cavernosa in order to theoretically provide a protective backing on the urethra.
  Interventions: Device: Artificial Urinary Sphincter
- Standard AUS (Active Comparator): The artificial urinary sphincter is placed in the standard fashion.
  Interventions: Device: Artificial Urinary Sphincter

INTERVENTIONS:
Device: Artificial Urinary Sphincter

SUMMARY:
We propose a randomized non-blinded comparison of standard vs. transcorporal approach for placement of an artificial urinary sphincter in male patients with stress urinary incontinence after radiation and radical prostatectomy for prostate cancer. In the United States, the artificial urinary sphincter (AUS), manufactured by American Medical Systems, is the gold standard surgical treatment for stress urinary incontinence (SUI) in men. The cuff, which is the portion of the device that encircles and occludes the urethra, is typically placed directly around the urethra (i.e., "standard" placement). The cuff can erode into the urethra. Transcorporal placement has been introduced as a method to reduce the risk of erosion. Transcorporal placement involves tunneling the cuff through the erectile bodies so as to protect the dorsal aspect of the urethra. This approach has never been compared to standard placement in a randomized fashion. In our randomized trial, no additional procedures beyond the normal care protocol will be required of the patients. We will conduct the study through our established, IRB-approved multi-institutional network of surgeons. Success will be assessed via objective and subjective methods; complications will be tallied in a standardized fashion. Outcomes will be measured at two years.

DETAILED DESCRIPTION:
The AUS is the gold standard for treatment of severe SUI, particularly in patients following surgical resection of the prostate for prostate cancer. In fact, severe urinary incontinence can be the most distressing complication following radical prostatectomy and results in a negative impact on quality of life (Haab, Trockman et al. 1997). Placement of an AUS has been shown to result in an improved quality of life in these patients. AUSs are small devices that prevent urinary flow via compression of the urethra, thus mimicking the native urinary sphincter. They have been available, albeit with occasional improvements or changes in design, since the 1970's. When placed in the standard fashion (ST) a small incision is made in the patient's perineum or scrotum and a fluid-filled cuff is placed around the bulbar urethra (the portion of the urethra between the bladder neck and penis). Connected to the cuff with tubing, is a balloon filled with fluid that is placed behind the pubic bone or in the space between the peritoneum and abdominal muscles. A control pump is placed in the scrotum and allows the device to cycle, thus either exerting pressure to close off the urethra or releasing pressure to allow the urethra to open and the patient to void. 73-76% of patients will experience dramatic improvement in incontinence with very minimal leakage (0-1 pads per day) and 88-89% report significant improvement or cure. Two years following implant, 9% of patients will experience a significant decline in the functionality of the device and report severe incontinence. At 5 years, 28% will need to undergo revision of the device (Dalkin, Wessells et al. 2003). Long-term complications associated with the device include urethral erosion in 5% of cases, urethral atrophy, infection, and mechanical failure of the device.

Patients undergoing radical prostatectomy frequently undergo radiation treatment during the course of their illness. Radiation to the pelvic region is responsible for compromising blood flow to the urethra and fibrosis. As a result these patients are at a moderate risk of developing complications and ultimately failure of the device necessitating removal and/or replacement. Factors that put patients in a high-risk category include a history of urethroplasty for urethral stricture, a history of a prior artificial urinary sphincter, and a history of open surgery for bladder neck contractures (scarring at the entrance to the bladder). Patients who develop a complication as listed above, often require a replacement AUS in a different location than the first cuff. This is done more distally in the penis where the urethra is narrower and there is less tissue to fill the cuff. This puts them at a higher risk for further complications. Several authors have recently published their experience with a modification to the standard technique in patients at a high risk for failure (Guralnick, Miller et al. 2002) (Aaronson, Elliott et al. 2008). The modified technique, termed transcorporal placement (TC), has been shown to be beneficial in this subset of patients. In one study, 28% of high-risk patients with ST placement developed erosion or infection, which required explanting the device compared with 13% in the TC group (4). Continence was also better in this high-risk group when TC placement was used, compared with ST, 89% vs 61%. TC placement also reduces the risk of injury to the urethra during surgery. Unlike in ST, TC placement involves placing the device around the urethra but also incorporating a flap of the tough tunica albigunea. The same incision is made as for the ST approach, and then an incision is made in each corpus cavernosum (cylinders of tissue that allow for erection). This allows the cuff to be placed around both the urethra and through the lining of the corporal bodies, increasing the bulk of tissue behind the urethra to protect it from erosion.

It has been suggested that placing the cuff near the erectile tissues might cause erectile dysfunction and as a result few surgeons perform this procedure on potent patients. However, scant data exist to support or refute this hypothetical effect on erectile function. Despite its success in patients at high risk of erosion, the TC approach has never been adequately tested in patients without a high risk of failure. It is unknown if this is a technique that only benefits this subset of patients or whether all patients might experience better long-term continence with less risk for erosion.

Study Objectives

The purpose of this study is to improve long-term patient outcomes and reduce complications and morbidity in patients with male SUI who are candidates for AUS insertion after radiation. The results from this study will provide clinicians evidence for superiority of either the ST or TC AUS. Our null hypothesis is that there is no difference in outcomes (as defined below) for AUS done in a TC vs. ST method. The alternative hypothesis is that one procedure is inferior/superior to the other.

Primary endpoint: AUS revision or removal surgery. These include surgery for mechanical failure, cuff erosion, impending erosion (discretion of surgeon), urethral atrophy, urinary incontinence and persistent retention due to small cuff.

Secondary endpoints:

Rate of post-operative urinary retention. Urinary retention defined as urinary catheter placement for more than 5 days in the period between AUS implantation and AUS activation (typically 4-8 weeks postoperatively) Incontinence at 3 months post-operatively measured using 24-hour pad weight test. Erectile function at 3 months as measured via the Sexual Health Inventory for Men (SHIM) Incontinence and QoL impact at 3 months as measured by the Incontinence Severity Index (ISI) and the Incontinency Impact Questionnaire Short From (IIQ-7)

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing an AUS procedure
* History of pelvic radiation for prostate or other cancer
* No spontaneous erections and no erections with oral erectogenic agents
* Subjects able to consent for themselves

Exclusion Criteria:

* prior urethroplasty
* prior urethral erosion of AUS
* history of penile prosthesis placement or explantation
* concomitant placement of penile prosthesis at the time of AUS placement

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
AUS Removal/Revision | 2 years
  We will record the incidence of any repeat AUS surgery for mechanical failure, cuff erosion, impending erosion (discretion of surgeon), urethral atrophy, urinary incontinence and persistent retention due to small cuff.

SECONDARY OUTCOMES:
Urinary Retention | 8 weeks
  Incidence of post-operative urinary retention defined as having a urethral catheter placed or re-placed any time after 5 days post-operative.
Incontinence | 3 months
  24 hour pad weight test will be administered at 3 months.
Incontinence Quality of Life | 3 months
  Incontinence Severity Index and Incontinency Impact Questionnaire Short Form questionnaire will be administered
Sexual Function | 3 months
  Sexual Health Inventory for Men will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Sean Elliott, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Aaronson DS, Elliott SP, McAninch JW. Transcorporal artificial urinary sphincter placement for incontinence in high-risk patients after treatment of prostate cancer. Urology. 2008 Oct;72(4):825-7. doi: 10.1016/j.urology.2008.06.065. Epub 2008 Aug 26. PMID 18752838
- [Background] Dalkin BL, Wessells H, Cui H. A national survey of urinary and health related quality of life outcomes in men with an artificial urinary sphincter for post-radical prostatectomy incontinence. J Urol. 2003 Jan;169(1):237-9. doi: 10.1016/S0022-5347(05)64076-1. PMID 12478144
- [Background] Guralnick ML, Miller E, Toh KL, Webster GD. Transcorporal artificial urinary sphincter cuff placement in cases requiring revision for erosion and urethral atrophy. J Urol. 2002 May;167(5):2075-8; discussion 2079. PMID 11956443
- [Background] Haab F, Trockman BA, Zimmern PE, Leach GE. Quality of life and continence assessment of the artificial urinary sphincter in men with minimum 3.5 years of followup. J Urol. 1997 Aug;158(2):435-9. PMID 9224318
- [Background] Simhan J, Morey AF, Zhao LC, Tausch TJ, Scott JF, Hudak SJ, Mazzarella BC. Decreasing need for artificial urinary sphincter revision surgery by precise cuff sizing in men with spongiosal atrophy. J Urol. 2014 Sep;192(3):798-803. doi: 10.1016/j.juro.2014.03.115. Epub 2014 Apr 16. PMID 24746880